CLINICAL TRIAL: NCT03848221
Title: Direct Application of Systane Complete to Contact Lenses for the Treatment of Contact Lens Discomfort
Brief Title: Direct Application of Systane Complete to Contact Lenses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Andrew Pucker, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 000523741
Record Dates: First submitted 2019-02-19; First posted 2019-02-20 (Actual); Results first posted 2020-04-27 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Dry Eye; Contact Lens Complication
Keywords: Systane Complete; Dry Eye; Contact Lens Discomfort; Artificial Tears; Rewetting Drops
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Investigator Masked, Randomized, Clinical Trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigator will be masked to the subject's treatment. The subjects cannot be fully masked because there is a no treatment control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Systane Complete (Experimental): Subjects in this group will use Systane Complete before, during, and after contact lens use.
  Interventions: Drug: Systane Complete
- Sensitive Eyes Rewetting Drops (Active Comparator): Subjects in this group will use Sensitive Eyes Rewetting Drops before, during, and after contact lens use.
  Interventions: Drug: Sensitive Eyes Rewetting Drops
- No Treatment (No Intervention): Subjects in this group will not be allowed to use artificial tears or rewetting drops during the study.

INTERVENTIONS:
Drug: Systane Complete — Systane Complete is an artificial tear.
  Arms: Systane Complete
Drug: Sensitive Eyes Rewetting Drops — Sensitive Eyes Rewetting Drops is a rewetting drop.
  Arms: Sensitive Eyes Rewetting Drops

SUMMARY:
A common first line treatment for patients with dryness symptoms or contact lens discomfort is the application of artificial tears or rewetting drops, respectively. Rewetting drops are specifically formulated for use with contact lenses while artificial tears are indicated for dry eye. Modern rewetting drops and artificial tears have similar formulations with similar preservatives, preservatives that have been shown to be compatible with contact lenses. While rewetting drops and artificial tears are regulated under different U.S. Food & Drug Administration policies, artificial tears are not specifically indicated for direct use with contact lenses. Nevertheless, clinicians commonly prescribe artificial tears to contact lens wearers likely because newer formulations of artificial tear have the potential to outperform available rewetting drops. The safety and efficacy of using artificial tears with contact lenses for the treatment of discomfort is supported by Caffery and Josephson and Ozkan and Papas who found that artificial tears significantly reduces dryness symptoms in contact lens wearers. Thus, the purpose of this study is to test the safety of directly applying a new artificial tear, Systane Complete, to the contact lens wearing eye and its ability to alleviate symptoms while wearing contact lenses during the day.

DETAILED DESCRIPTION:
Soft contact lenses are the ideal vision correction choice for many patients because soft contact lenses allow patients to have better and less restricted vision, they allow for an increased ability to perform work tasks and play sports, and they provide patients with a better perceived cosmetic appearance compared to spectacle lenses. While millions of people worldwide benefit from contact lenses, many of these patients experience contact lens discomfort, which limits their wear time and in many instances eventually result in discontinuation of contact lens use. In fact, 21% to 64% of contact lens wearers permanently discontinue contact lens use because of ocular discomfort. Contact lens discomfort is currently defined as "a condition characterized by episodic or persistent adverse ocular sensations related to lens wear, either with or without visual disturbance, resulting from reduced compatibility between the contact lens and the ocular environment, which can lead to decreased wearing time and discontinuation of contact lens wear." Although contact lens discomfort may stem from the lens itself, a situation that can be corrected by such means as switching to an alternative material or wear schedule, contact lens discomfort more typically occurs from ocular surface disease.

A common first line treatment for patients with dryness symptoms or contact lens discomfort is the application of artificial tears or rewetting drops, respectively. Rewetting drops are specifically formulated for use with contact lenses while artificial tears are indicated for dry eye. Modern rewetting drops and artificial tears have similar formulations with similar preservatives, preservatives that have been shown to be compatible with contact lens use. While rewetting drops and artificial tears are regulated under different U.S. Food & Drug Administration policies, artificial tears are not specifically indicated for use with contact lenses. Nevertheless, clinicians commonly prescribe artificial tears to contact lens wearers likely because newer formulations of artificial tear have the potential to outperform available rewetting drops (e.g., some artificial tears have lipid supplements that have the potential to restore the external tear lipid layer). The safe and effective use of artificial tears with contact lenses is supported by Caffery and Josephson and Ozkan and Papas who found that artificial tears significantly reduce dryness symptoms in contact lens wearers. However, the community currently lacks a rigorous scientific study aimed at understanding the utility of lipid-containing artificial tear (or rewetting drop) for alleviating contact lens discomfort while patients are wearing their contact lenses. Systane Complete, a new formulation of artificial tears, combines elements from both Systane Ultra (indicated for aqueous deficient dry eye) and Systane Balance (lipid-containing artificial tear indicated for evaporative dry eye). Thus, the purpose of this study is to test the safety of Systane Complete and its ability to alleviate contact lens discomfort during the day while subjects are wearing their contact lenses. This goal will be accomplished by randomizing subjects to either Systane Complete, a commercially available rewetting drop, or no treatment.

ELIGIBILITY:
Inclusion Criteria:

* Daily disposable contact lens wearers
* 20/30 visual acuity or better
* Self-report contact lens discomfort
* Contact Lens Dry Eye Questionnaire (CLDEQ)-8 scores ≥ 12

Exclusion Criteria:

* Other contact lens modalities/wear schedules (e.g., two week and monthly replacement CLs, gas permeable CLs)
* Non-compliant daily disposable contact lens wearers
* Systemic health conditions that alter tear film physiology (e.g., primary and secondary Sjögren's syndrome)
* History of ocular surgery within the past 12 months
* History of severe ocular trauma
* History of active ocular infection or inflammation
* Isotretinoin-derivatives use
* Ocular medication use
* Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2019-10-20 (Actual); Study Completion 2019-10-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Lindenhurst Eye Physicians & Surgeons, P.C., Babylon, New York
  - Southern College of Optometry, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual subject data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Systane Complete | Sensitive Eyes Rewetting Drops | No Treatment
Started | 25 | 24 | 24
Completed | 25 | 24 | 24
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects were included if they were generally healthy adult (18 years or older) contact lens wearer who had significant contact lens and dry eye questionnaire cldeq8 scores of 12 or greater.
Groups:
- Total: Total of all reporting groups
Arm/Group | Systane Complete | Sensitive Eyes Rewetting Drops | No Treatment | Total
Number analyzed (Participants) | 25 | 24 | 24 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 24 | 24 | 73
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 20 | 60
  Male | 4 | 5 | 4 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 24 | 73

OUTCOME MEASURES:

1. Primary Outcome: Difference in Ocular Surface Damage as Measured by the Brien Holden Vision Institute (BHVI Grading Scale) at Two Weeks
Description: The Corneal Staining Scores are measured by the BHVI grading scale. The grading scales are a quick reference to the key signs associated with contact lens related inflammation and infection. Used as a reference tool in the clinic, they provide a guide for determining how much normal ocular appearance has changed in a patient, and can help inform clinical management decisions. The range of the scores are: 0-4 in five regions (total sum score = 20). A lower score indicates a better outcome.
Time Frame: 2 Weeks
Population: Generally healthy adults who had a significant CLDEQ-8 score and were contact lens wearers.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Systane Complete | Sensitive Eyes Rewetting Drops | No Treatment
Number analyzed (Participants) | 25 | 24 | 24
Score on a Scale | 0.44 (0.82) | 1.08 (1.32) | 0.83 (1.99)
Statistical Analysis 1: Comparison: Systane Complete vs Sensitive Eyes Rewetting Drops vs No Treatment; Test type: Equivalence; p = 0.30, ANOVA

2. Secondary Outcome: Identifying Contact Lens (CL) Participants With Dry Eye Disease (DED), as Measured by the Contact Lens Dry Eye Questionnaire-4 Items (CLDEQ-4) Between Two Weeks and Baseline.
Description: The CLDEQ-4 is a contact lens specific symptoms survey; range = 0-18 with 18 being most symptomatic.
Time Frame: 2 Weeks
Population: Generally healthy adults who had a significant CLDEQ-8 score and were contact lens wearers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Systane Complete | Sensitive Eyes Rewetting Drops | No Treatment
Number analyzed (Participants) | 25 | 24 | 24
score on a scale | -8.52 (2.97) | -8.25 (2.42) | -11.50 (3.08)
Statistical Analysis 1: Comparison: Systane Complete vs Sensitive Eyes Rewetting Drops vs No Treatment; Test type: Equivalence; p = 0.0002, ANOVA

ADVERSE EVENTS:
Time Frame: Two Weeks.
Arm/Group | Systane Complete | Sensitive Eyes Rewetting Drops | No Treatment
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT03848221/Prot_SAP_ICF_002.pdf